CLINICAL TRIAL: NCT02638818
Title: A Pilot Study Evaluating Health-related Quality of Life Endpoints in Patients Undergoing Minimally Invasive Versus Open Pancreaticoduodenectomy
Brief Title: Outcomes in Minimally Invasive Versus Open Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00064629
Record Dates: First submitted 2015-11-30; First posted 2015-12-23 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Disease
Keywords: pancreaticoduodenectomy; Whipple
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- minimally invasive whipple: Surgical technique (minimally invasive vs open) will be at the discretion of the operating surgeon. Patients will not be randomized to a treatment arm.
  Interventions: Procedure: minimally invasive pancreaticoduodenectomy
- traditional whipple: Surgical technique (minimally invasive versus open) will be at the discretion of the operating surgeon. Patients will not be randomized to a treatment arm.
  Interventions: Procedure: traditional pancreaticoduodenectomy

INTERVENTIONS:
Procedure: minimally invasive pancreaticoduodenectomy — Surgical technique (minimally invasive versus open) will be at the discretion of the operating surgeon. Patients will not be randomized to a treatment arm.
  Groups: minimally invasive whipple
Procedure: traditional pancreaticoduodenectomy — Surgical technique (minimally invasive versus open) will be at the discretion of the operating surgeon. Patients will not be randomized to a treatment arm.
  Groups: traditional whipple

SUMMARY:
The purpose of this study is to evaluate the impact of the quality of life in patients undergoing the Whipple procedure (pancreaticoduodenectomy, PD) for pancreatic cancer. The Whipple procedure can be done by laparoscopic (small incisions) or an open procedure (large incision) to treat the patients cancer. The goal of this study is to see if there is any difference in quality of life between patients who undergo the laparoscopic or the open Whipple procedure. Surgical technique (minimally invasive versus open) will be at the discretion of the operating surgeon. Patients will not be randomized to a treatment arm.

A subset of these patients will also be asked to take part in a pre- and postoperative in-depth interview to explore the lived experiences of patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for pancreaticoduodenectomy will be eligible for this study.
* Subject must be at least 18 years of age and at least the minimum Age of Majority according to applicable State or Country Law.
* Subject is a suitable surgical candidate, i.e. is able to undergo general anesthesia and PD for diagnosis of cancer
* Subject is willing and able to cooperate with survey participation.
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form

Exclusion Criteria:

• Subject is not a suitable candidate for PD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for pancreaticoduodenectomy will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Change in quality of life, as measured by FACT-Hep score | Baseline (before surgery), at hospital discharge (up to approximately 14 days), at first clinic visit (within 2 weeks after discharge), 3 months
  The summed overall FACT-Hep score (0-180) will be the primary outcome.

IPD SHARING:
Plan to Share IPD: Undecided